CLINICAL TRIAL: NCT03614221
Title: Comparison of the Efficacy and Safety of Lindioil (Indigo Naturalis Oil Extract) Ointment to Protopic® (Tacrolimus 0.1%) Ointment in Treating Atopic Dermatitis: A Randomized, Evaluator-blind, Crossover, Active-Controlled Trial
Brief Title: Comparison of Lindioil (Indigo Naturalis Oil Extract) Ointment to Protopic® Ointment 0.1% in Treating Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MOST107-2320-B-182A-002 -MY3
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Indigo naturalis; Tacrolimus
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lindioil (Experimental): Lindioil ointment is applied twice daily for 6 weeks, followed by a washout period of 4 days to 8 weeks depending on the results of the first treatment period and the amount of time it takes the participant to relapse to IGA ≥ 2 and less than 1-point of change from baseline1ST IGA. If relapse to IGA ≥ 2 and less than 1-point of change from baseline1ST IGA is achieved, the patient is using Protopic ointment 0.1% twice daily for another 6 weeks. If the criteria for entering the 2nd treatment are not achievable after 8-week of ceasing 1st treatment, the subject will be followed up for another 6 weeks to the end of the study
  Interventions: Drug: Lindioil ointment; Drug: Protopic ointment 0.1%
- Protopic (Active Comparator): Protopic ointment 0.1% is applied twice daily for 6 weeks, followed by a washout period of 4 days to 8 weeks depending on the results of the first treatment period and the amount of time it takes the participant to relapse to IGA ≥ 2 and less than 1-point of change from baseline1ST IGA. If relapse to IGA ≥ 2 and less than 1-point of change from baseline1ST IGA is achieved, the patient is using Lindioil ointment twice daily for another 6 weeks. If the criteria for entering the 2nd treatment are not achievable after 8-week of ceasing 1st treatment, the subject will be followed up for another 6 weeks to the end of the study
  Interventions: Drug: Lindioil ointment; Drug: Protopic ointment 0.1%

INTERVENTIONS:
Drug: Lindioil ointment — Each gram contains 200µg of indirubin. Apply 0.5 g of ointment per 10 cm x 10 cm of affected skin areas twice daily for 6 weeks.
  Other Names: Indigo naturalis oil extract ointment
Drug: Protopic ointment 0.1% — Each gram contains (w/w) 0.1% of tacrolimus. Apply 0.1 g of ointment per 10 cm x 10 cm of affected skin areas twice daily for 6 weeks.
  Other Names: Tacrolimus ointment 0.1%

SUMMARY:
The aims of this study are:

1. Compare the efficacy of Lindioil ointment and Protopic® ointment in treating atopic dermatitis.
2. Compare the safety of Lindioil ointment and Protopic® ointment in treating atopic dermatitis.
3. Compare the time to relapse after ceasing of treatment of Lindioil ointment and Protopic® ointment.
4. Compare the change of skin microbiome before and after Lindioil ointment and Protopic® ointment treatment.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory skin disorder characterized by itchiness. Topical corticosteroids are typically used to treat AD. However, many patients have concerns about the safety of long-term use, and seek alternative therapies such as traditional Chinese medicine (TCM). In TCM, indigo naturalis has been used to treat various infectious and inflammatory skin diseases for hundreds of years. The investigate also found that the results of indigo naturalis ointment treatment in other trial were comparable to the results of calcineurin inhibitor (such as Tacrolimus) treatment, and would like to verify this assertion. The aim of this study is to compare the efficacy of Lindioil ointment with that of Protopic® (Tacrolimus ointment 0.1%) in treating AD.

ELIGIBILITY:
Inclusion Criteria:

1. Between 16 and 65 years old, female or male.
2. Chronic or sub-acute atopic dermatitis fulfilling the United Kingdom (UK) diagnostic criteria of atopic dermatitis.
3. Atopic dermatitis involving 3-40% of BSA at screening and baseline.
4. An IGA score of 2 (mild) to 4 (severe) at screening and baseline.
5. Not supposed to or unwilling to use corticosteroids.
6. Female patients of child-bearing age agree to use effective birth control measures approved by the investigator.
7. Agree to avoid natural and artificial sunlight over-exposure during the study.
8. Willing to comply with study protocol and agree to sign an informed consent form

Exclusion Criteria:

1. Acute atopic dermatitis or concurrence of viral or bacterial infection on dermatitis lesion(s).
2. A history of topical or systematic hypersensitivity to indigo naturalis, tacrolimus, or the excipient(s) in the ointment(s).
3. Having received systemic therapy (e.g. immunosuppressive agents) within 14 days, or phototherapy (e.g.

   ultraviolet B (UVB), psoralen and ultraviolet A (PUVA)) within 42 days before the first application of the study medication.
4. Having used topical therapy (e.g. corticosteroids) for dermatitis within 4 days before the first application of the study medication.
5. Having a significant concurrent disease such as severe uncontrolled chronic disease (e.g., hypertension, diabetes mellitus, metabolic arthritis, hyperthyroidism), psychiatric disease, cancer or AIDS.
6. Having significant abnormal liver or renal function (Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) >3 x upper limit of normal (ULN), creatinine >2.0 mg/dl) or clinically significant abnormal hematological lab result, according to investigator's judgment, on the safety lab test to be performed within 30 days before the baseline visit.
7. Women who are lactating, pregnant or planning to be pregnant during the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
The mean percentage change from baseline to the end of week 6 of Eczema Area Severity Index (EASI) scores (range 0-72), for each of the two 6-week treatment periods. | 6-week, 12-week (the end of the second treatment period)
  The Eczema Area and Severity Index (EASI) is used to measure the disease severity of erythema, infiltration/papulation, excoriation, and lichenification each on a scale of 0 to 3 (none to severe) as well as the percentage of disease area on a scale of 0 to 6 for the 4 body regions: head ⁄ neck, upper limbs, trunk and lower limbs. Each body region score is calculated by multiplying the disease severity score by the disease area score and by the multiplier, 0.1 for head/neck, 0.2 for upper limbs, 0.3 for trunk, and 0.4 for lower limbs. The scores are summed to give the total EASI score, ranging from 0 to a maximum 72.

SECONDARY OUTCOMES:
Proportion of participants who have achieved a 50%, 75% and 90% improvement in EASI scores (EASI-50, EASI-75 and EASI-90, respectively) at the end of week 6 of each treatment period. | 6-week, 12-week (the end of the second treatment period)
  It is defined as at least 50%, 75%, and 90% reduction in EASI score compare to the baseline.
Proportion of participants with an Investigator's Global Assessment (IGA, 0-5) score of 0 (clear) or 1 (almost clear) at the end of week 6 of each treatment period. | 6-week, 12-week (the end of the second treatment period)
  Investigator's Global Assessment (IGA) is a 6-points scale ranging from 0 (cleared) to 5 (Very severe) for evaluation of the severity of atopic dermatitis.
The mean percentage change from baseline to the end of week 6 of the Body Surface Area (BSA, range 0%-100%) affected by AD, for each of the two 6-week treatment periods. | 6-week, 12-week (the end of the second treatment period)
  BSA is total body surface area affected by atopic dermatitis, ranging from 0% (none) to 100% (total body surface affected).
Number of days until relapse to IGA ≥ 2, after ceasing treatment, for subjects who achieved IGA 0 or 1 at the end of week 6 of each treatment period. | 6-week, 12-week (the end of the second treatment period)
  Length of relapse free days after ceasing treatment
The change from baseline to the end of week 6 of Numeric Rating Scale for pruritus (NRS, 0-10), for each of the two 6-week treatment periods. | 6-week, 12-week (the end of the second treatment period)
  Numeric Rating Scale for pruritus (NRS) is a tool to evaluate itching intensity from 0 (no itch) to 10 (most imaginable itch)
The change from baseline to the end of week 6 of Dermatology Life Quality Index (DLQI) for each of the two 6-week treatment periods. | 6-week, 12-week (the end of the second treatment period)
  The DLQI is a self-administered 10-item questionnaire, ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.
Proportion of participants with a Subject's Global Assessment (SGA, 0-6) score of 0 (much better) or 1 (better) at the end of week 6 of each treatment period. | 6-week, 12-week (the end of the second treatment period)
  Subject's Global Assessment (SGA) is a self-evaluated the change from baseline of their AD condition as 'much better' (0), 'better' (1) , 'slightly better' (2), 'same' (3), 'slightly worse' (4), 'worse' (5) or 'much worse' (6).
The participants' preference of using Lindioil ointment and Protopic® ointment treatment. | 13 weeks (the end of the second treatment period)
  Patients who completed the second treatment period will answer which ointment with better efficacy, which with more adverse events, and the adverse event bothering them most.
The change of skin microbiome before and after Lindioil ointment and Protopic® ointment treatment. | 6-week, 12-week (the end of the second treatment period)
  Skin swabs of lesion and non-lesion will be obtained from patient before and after study treatment to analyze skin microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ku Lin, MD., PhD., Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Taipei Chang Gung Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Background] Al-Daraji WI, Grant KR, Ryan K, Saxton A, Reynolds NJ. Localization of calcineurin/NFAT in human skin and psoriasis and inhibition of calcineurin/NFAT activation in human keratinocytes by cyclosporin A. J Invest Dermatol. 2002 May;118(5):779-88. doi: 10.1046/j.1523-1747.2002.01709.x. PMID 11982754
- [Background] Caproni M, Torchia D, Antiga E, Terranova M, Volpi W, del Bianco E, D'Agata A, Fabbri P. The comparative effects of tacrolimus and hydrocortisone in adult atopic dermatitis: an immunohistochemical study. Br J Dermatol. 2007 Feb;156(2):312-9. doi: 10.1111/j.1365-2133.2006.07609.x. PMID 17223872
- [Background] Simon D, Vassina E, Yousefi S, Kozlowski E, Braathen LR, Simon HU. Reduced dermal infiltration of cytokine-expressing inflammatory cells in atopic dermatitis after short-term topical tacrolimus treatment. J Allergy Clin Immunol. 2004 Oct;114(4):887-95. doi: 10.1016/j.jaci.2004.05.066. PMID 15480330
- [Background] Furukawa H, Nakamura K, Zheng X, Tojo M, Oyama N, Akiba H, Nishibu A, Kaneko F, Tsunemi Y, Saeki H, Tamaki K. Enhanced TARC production by dust-mite allergens and its modulation by immunosuppressive drugs in PBMCs from patients with atopic dermatitis. J Dermatol Sci. 2004 Jun;35(1):35-42. doi: 10.1016/j.jdermsci.2004.02.008. PMID 15194145
- [Background] Chang KT, Lin HY, Kuo CH, Hung CH. Tacrolimus suppresses atopic dermatitis-associated cytokines and chemokines in monocytes. J Microbiol Immunol Infect. 2016 Jun;49(3):409-16. doi: 10.1016/j.jmii.2014.07.006. Epub 2014 Oct 12. PMID 25315214
- [Background] Vukmanovic-Stejic M, McQuaid A, Birch KE, Reed JR, Macgregor C, Rustin MH, Akbar AN. Relative impact of CD4+CD25+ regulatory T cells and tacrolimus on inhibition of T-cell proliferation in patients with atopic dermatitis. Br J Dermatol. 2005 Oct;153(4):750-7. doi: 10.1111/j.1365-2133.2005.06675.x. PMID 16181456
- [Background] Lan CC, Kao YH, Huang SM, Yu HS, Chen GS. FK506 independently upregulates transforming growth factor beta and downregulates inducible nitric oxide synthase in cultured human keratinocytes: possible mechanisms of how tacrolimus ointment interacts with atopic skin. Br J Dermatol. 2004 Sep;151(3):679-84. doi: 10.1111/j.1365-2133.2004.06109.x. PMID 15377358
- [Background] Paller AS, Lebwohl M, Fleischer AB Jr, Antaya R, Langley RG, Kirsner RS, Blum RR, Rico MJ, Jaracz E, Crowe A, Linowski GJ; US/Canada Tacrolimus Ointment Study Group. Tacrolimus ointment is more effective than pimecrolimus cream with a similar safety profile in the treatment of atopic dermatitis: results from 3 randomized, comparative studies. J Am Acad Dermatol. 2005 May;52(5):810-22. doi: 10.1016/j.jaad.2004.12.038. PMID 15858471
- [Background] Breneman D, Fleischer AB Jr, Abramovits W, Zeichner J, Gold MH, Kirsner RS, Shull TF, Crowe AW, Jaracz E, Hanifin JM; Tacrolimus Ointment Study Group. Intermittent therapy for flare prevention and long-term disease control in stabilized atopic dermatitis: a randomized comparison of 3-times-weekly applications of tacrolimus ointment versus vehicle. J Am Acad Dermatol. 2008 Jun;58(6):990-9. doi: 10.1016/j.jaad.2008.02.008. Epub 2008 Mar 21. PMID 18359127
- [Background] Lin YK, Chang CJ, Chang YC, Wong WR, Chang SC, Pang JH. Clinical assessment of patients with recalcitrant psoriasis in a randomized, observer-blind, vehicle-controlled trial using indigo naturalis. Arch Dermatol. 2008 Nov;144(11):1457-64. doi: 10.1001/archderm.144.11.1457. PMID 19015420
- [Background] Lin YK, Chang YC, Hui RC, See LC, Chang CJ, Yang CH, Huang YH. A Chinese Herb, Indigo Naturalis, Extracted in Oil (Lindioil) Used Topically to Treat Psoriatic Nails: A Randomized Clinical Trial. JAMA Dermatol. 2015 Jun;151(6):672-4. doi: 10.1001/jamadermatol.2014.5460. No abstract available. PMID 25738921
- [Background] Lin YK, See LC, Huang YH, Chang YC, Tsou TC, Lin TY, Lin NL. Efficacy and safety of Indigo naturalis extract in oil (Lindioil) in treating nail psoriasis: a randomized, observer-blind, vehicle-controlled trial. Phytomedicine. 2014 Jun 15;21(7):1015-20. doi: 10.1016/j.phymed.2014.02.013. Epub 2014 Mar 26. PMID 24680615
- [Background] Lin YK, See LC, Huang YH, Chi CC, Hui RC. Comparison of indirubin concentrations in indigo naturalis ointment for psoriasis treatment: a randomized, double-blind, dosage-controlled trial. Br J Dermatol. 2018 Jan;178(1):124-131. doi: 10.1111/bjd.15894. Epub 2017 Dec 14. PMID 28815560
- [Background] Hoessel R, Leclerc S, Endicott JA, Nobel ME, Lawrie A, Tunnah P, Leost M, Damiens E, Marie D, Marko D, Niederberger E, Tang W, Eisenbrand G, Meijer L. Indirubin, the active constituent of a Chinese antileukaemia medicine, inhibits cyclin-dependent kinases. Nat Cell Biol. 1999 May;1(1):60-7. doi: 10.1038/9035. PMID 10559866
- [Background] Marko D, Schatzle S, Friedel A, Genzlinger A, Zankl H, Meijer L, Eisenbrand G. Inhibition of cyclin-dependent kinase 1 (CDK1) by indirubin derivatives in human tumour cells. Br J Cancer. 2001 Jan;84(2):283-9. doi: 10.1054/bjoc.2000.1546. PMID 11161389
- [Background] Sethi G, Ahn KS, Sandur SK, Lin X, Chaturvedi MM, Aggarwal BB. Indirubin enhances tumor necrosis factor-induced apoptosis through modulation of nuclear factor-kappa B signaling pathway. J Biol Chem. 2006 Aug 18;281(33):23425-35. doi: 10.1074/jbc.M602627200. Epub 2006 Jun 19. PMID 16785236
- [Background] Kunikata T, Tatefuji T, Aga H, Iwaki K, Ikeda M, Kurimoto M. Indirubin inhibits inflammatory reactions in delayed-type hypersensitivity. Eur J Pharmacol. 2000 Dec 20;410(1):93-100. doi: 10.1016/s0014-2999(00)00879-7. PMID 11134660
- [Background] Cheng HM, Wu YC, Wang Q, Song M, Wu J, Chen D, Li K, Wadman E, Kao ST, Li TC, Leon F, Hayden K, Brodmerkel C, Chris Huang C. Clinical efficacy and IL-17 targeting mechanism of Indigo naturalis as a topical agent in moderate psoriasis. BMC Complement Altern Med. 2017 Sep 2;17(1):439. doi: 10.1186/s12906-017-1947-1. PMID 28865459
- [Background] Lin YK, Chen HW, Leu YL, Yang YL, Fang Y, Su Pang JH, Hwang TL. Indigo naturalis upregulates claudin-1 expression in human keratinocytes and psoriatic lesions. J Ethnopharmacol. 2013 Jan 30;145(2):614-20. doi: 10.1016/j.jep.2012.11.044. Epub 2012 Dec 7. PMID 23220199
- [Background] Lin YK, Leu YL, Yang SH, Chen HW, Wang CT, Pang JH. Anti-psoriatic effects of indigo naturalis on the proliferation and differentiation of keratinocytes with indirubin as the active component. J Dermatol Sci. 2009 Jun;54(3):168-74. doi: 10.1016/j.jdermsci.2009.02.007. Epub 2009 Mar 19. PMID 19303259
- [Background] Chang HN, Pang JH, Yang SH, Hung CF, Chiang CH, Lin TY, Lin YK. Inhibitory effect of indigo naturalis on tumor necrosis factor-alpha-induced vascular cell adhesion molecule-1 expression in human umbilical vein endothelial cells. Molecules. 2010 Sep 14;15(9):6423-35. doi: 10.3390/molecules15096423. PMID 20877233
- [Background] Chiang YR, Li A, Leu YL, Fang JY, Lin YK. An in vitro study of the antimicrobial effects of indigo naturalis prepared from Strobilanthes formosanus Moore. Molecules. 2013 Nov 21;18(11):14381-96. doi: 10.3390/molecules181114381. PMID 24284490
- [Background] Lin YK, Chen HW, Yang SH, Leu YL, Huang YH, Yen HC. Protective effect of indigo naturalis extract against oxidative stress in cultured human keratinocytes. J Ethnopharmacol. 2012 Feb 15;139(3):893-6. doi: 10.1016/j.jep.2011.12.037. Epub 2011 Dec 27. PMID 22212506
- [Background] Lin YK, Leu YL, Huang TH, Wu YH, Chung PJ, Su Pang JH, Hwang TL. Anti-inflammatory effects of the extract of indigo naturalis in human neutrophils. J Ethnopharmacol. 2009 Aug 17;125(1):51-8. doi: 10.1016/j.jep.2009.06.014. Epub 2009 Jun 25. PMID 19559779
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] Reitamo S, Ortonne JP, Sand C, Cambazard F, Bieber T, Folster-Holst R, Vena G, Bos JD, Fabbri P, Groenhoej Larsen C; European Tacrolimus Ointment Study Group. A multicentre, randomized, double-blind, controlled study of long-term treatment with 0.1% tacrolimus ointment in adults with moderate to severe atopic dermatitis. Br J Dermatol. 2005 Jun;152(6):1282-9. doi: 10.1111/j.1365-2133.2005.06592.x. PMID 15948994
- [Background] Byrd AL, Deming C, Cassidy SKB, Harrison OJ, Ng WI, Conlan S; NISC Comparative Sequencing Program; Belkaid Y, Segre JA, Kong HH. Staphylococcus aureus and Staphylococcus epidermidis strain diversity underlying pediatric atopic dermatitis. Sci Transl Med. 2017 Jul 5;9(397):eaal4651. doi: 10.1126/scitranslmed.aal4651. PMID 28679656
- [Background] Meylan P, Lang C, Mermoud S, Johannsen A, Norrenberg S, Hohl D, Vial Y, Prod'hom G, Greub G, Kypriotou M, Christen-Zaech S. Skin Colonization by Staphylococcus aureus Precedes the Clinical Diagnosis of Atopic Dermatitis in Infancy. J Invest Dermatol. 2017 Dec;137(12):2497-2504. doi: 10.1016/j.jid.2017.07.834. Epub 2017 Aug 24. PMID 28842320
- [Background] Fukushima H, Hirano T, Shibayama N, Miwa K, Ito T, Saito M, Sumida H, Oyake S, Tsuboi R, Oka K. The role of immune response to Staphylococcus aureus superantigens and disease severity in relation to the sensitivity to tacrolimus in atopic dermatitis. Int Arch Allergy Immunol. 2006;141(3):281-9. doi: 10.1159/000095298. Epub 2006 Aug 23. PMID 16931890
- [Derived] Yang CY, Chen CB, Lu CW, Chi MH, Wu J, Chung WH, Lee BH, Lin YK. Efficacy and safety of indigo naturalis oil extract (Lindioil ointment) for the treatment of atopic dermatitis: a randomized, crossover, evaluator-blinded, controlled trial. Front Pharmacol. 2025 Jul 8;16:1546589. doi: 10.3389/fphar.2025.1546589. eCollection 2025. PMID 40697652